CLINICAL TRIAL: NCT02292290
Title: A Randomised Controlled Trial for People With Established Type 2 Diabetes During Ramadan: Liraglutide vs. a Sulphonylurea
Brief Title: Trial for People With Established Type 2 Diabetes During Ramadan
Acronym: T4R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0207
Record Dates: First submitted 2011-01-16; First posted 2014-11-17 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2012-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Liraglutide; Ramadan; fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Fasting | interventions — Liraglutide; Sulfonylurea Compounds; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Monotherapy 2 (Active Comparator): addition of Sulfonylurea or Pioglitazone to Metformin
  Interventions: Drug: Sulfonylurea or Pioglitazone
- Dual Therapy 1 (Experimental): Swap Liraglutide for sulfonylurea or pioglitazone taken as second line therapy (Metformin) first line)
  Interventions: Drug: Liraglutide
- Dual therapy 2 (Active Comparator): Maintain sulfonylurea or pioglitazone as second line therapy (Metformin first line)
  Interventions: Drug: Maintain dual therapy (Sulf/Pio) as comparator to Liraglutide
- Monotherapy (Experimental): Addition of Liraglutide to Metformin
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — 4 week lead-in 0.6mg Liraglutide OD up to 1.2mg OD after 2 weeks if poor response
  Other Names: Victoza
  Arms: Monotherapy
Drug: Liraglutide — 4 week lead-in 0.6mg Liraglutide OD up to 1.2mg after two weeks if poor response.
  Other Names: Victoza
  Arms: Dual Therapy 1
Drug: Sulfonylurea or Pioglitazone — Addition to Metformin
  Arms: Monotherapy 2
Drug: Maintain dual therapy (Sulf/Pio) as comparator to Liraglutide — As per clinical guidelines for prescription
  Arms: Dual therapy 2

SUMMARY:
Dual therapy with metformin and Liraglutide is more effective at helping people with established Type 2 Diabetes Mellitus (T2DM) observing Ramadan achieve a triple composite endpoint of weight reduction and/or maintenance and improved HaemaglobinA1c (HbA1c) and no severe hypoglycaemic events.

DETAILED DESCRIPTION:
Participants in the control arm will essentially continue with their standard routine care and those in the intervention groups will either receive Liraglutide in addition to metformin or those on dual therapy will switch from their sulphonylurea/pioglitazone to Liraglutide and continue with metformin. Informed consent and baseline data will be collected 4-8 weeks prior to the start of Ramadan. This will allow time for a run in period for the titration of Liraglutide prior to the fasting period. Ramadan is followed by Eid-al-Fitr a 3-day Islamic holiday that marks the end of this holy month. Tradition includes amongst early morning prayers/celebration through feasting. Therefore, participants will be invited to attend the first follow-up after this event (between weeks 2 - 4) and then at 12 weeks post Ramadan. Randomisation will not be revealed until after the baseline data have been collected.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years old with established T2DM on metformin only
* or dual therapy of metformin plus a sulphonylurea or pioglitazone
* with a HbA1c between 7 - 11 % if on monotherapy and between 6.5 - 12% if on dual therapy

Exclusion Criteria:

* Are pregnant or breast feeding
* Suffer from terminal illness
* Have significant renal or liver impairment
* Are unable to provide informed consent
* Have severe and enduring mental health problems
* Are not primarily responsible for their own care
* Are receiving insulin therapy
* Type 1 diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Composite | 12 weeks following post Ramadan cinical assessment
  A composite endpoint of a reduction in weight, reduction/maintenance of HbA1c and elimination of severe hypoglycaemic (defined as hospital admission) events post intervention.

SECONDARY OUTCOMES:
HbA1c only | same as primary, 12 weeks following post Ramadan cinical assessment
  Mean change HbA1c level

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J D, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester, Leicester, Leicestershire
  - University Hospital Birmingham, Birmingham, West Midlands